CLINICAL TRIAL: NCT00359229
Title: A Multicentre Prospective, Open Label ,3 Weeks Phase IV Study to Evaluate the Efficacy and Safety in Elder Patients With Insomnia in China
Brief Title: Stilnox Treatment in Elderly Patients With Insomnia
Acronym: STEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZOLPI_L_01540
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

ARMS (1):
- 1 (Experimental): For 3 weeks
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: Zolpidem — Administration of Zolpidem 5mg

SUMMARY:
Primary objective:

1. To evaluate the efficacy of Zolpidem 5mg for 1 week in elderly patients with insomnia in China

Secondary objectives:

1. To evaluate the safety of Zolpidem 5mg for 3 weeks in elderly patients with insomnia in China.
2. To evaluate the efficacy of Zolpidem 5mg for 3 weeks in elderly patients with insomnia in China

ELIGIBILITY:
Inclusion Criteria:

* Primary out-patient insomniac patient defined by DSM-IV criteria
* Insomnia history lasted at least 3 months , this history must include a self-reported usual sleep latency of 30 minutes or more and either 3 or more awakenings per night on average or a usual total sleep time of ≤6.5 hours

Exclusion Criteria:

* Usage of hypnotics within the previous 1-3 weeks before inclusion depending on the half-life of the hypnotics that would affect the study effect
* Concomitant usage of other hypnotics (benzodiazepines and Non-benzodiazepines) during the course if the study.
* Concomitant usage of the following Central Nervous System active medicine : antipsychotics , antidepressants ,anxiolytics, lithium and other psychotropic drugs.
* The score of Hamilton Depression Rating Scale (HAMD-24 ) more than 17.
* The score of Hamilton Anxiety Rating Scale (HAMA-14 ) more than 14.
* Patients having known hypersensitivity to Stilnox or any of the ingredients in the products
* Patient with severe respiratory insufficiency
* Patients suffering from sleep apnoea syndrome
* Patients with known severe hepatic (risk of encephalopathy) and /or renal insufficiency, or other severe organ diseases
* Patients suffering from severe myasthenia gravis
* Patients with the previous history of drug abuse, drug dependence and drug addiction
* Any other disease state or major psychiatric condition that might affect study result

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) score | At 1 week versus baseline

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index score | At 3 weeks versus baseline
Subject sleeping efficacy variable | At 1 week and 3 weeks versus baseline
Hamilton Depression Rating Scale (HAMD) and Hamilton Anxiety Rating Scale (HAMA) score | At 3 weeks versus baseline
Adverse events (AE) and Serious adverse events (SAE) reports | Throughout the study period
General Lab tests including hepatic and renal function | At 3 weeks versus baseline
Vital signs | At 1 week and 3 weeks versus baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Jolain, Study Director — Sanofi